CLINICAL TRIAL: NCT05738083
Title: Multi-Center Registry Cohort Study on Prognostic Factors and Prediction Model Construction in Aneurysmal Subarachnoid Hemorrhage
Brief Title: Multi-Center Registry Cohort Study on Prognostic Factors and Prediction Model Construction in Aneurysmal SAH
Acronym: PROSAH-MPC
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Panzhihua Central Hospital (Other); Zhujiang Hospital (Other); Southwest Hospital, China (Other); Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-O-2023-011
Record Dates: First submitted 2022-11-16; First posted 2023-02-21 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- aneurysmal subarachnoid hemorrhage: primary subarachnoid hemorrhage caused by intracranial ruputured aneurysm
  Interventions: Diagnostic Test: Machine Leaning Models

INTERVENTIONS:
Diagnostic Test: Machine Leaning Models — Area Under the Curve (ROC): Measures the overall performance of the model across all classification thresholds. A higher AUC value indicates better performance.
  Accuracy: The proportion of correctly predicted outcomes (both positive and negative) out of all predictions made.
  Precision (Positive Predictive Value, PPV): The proportion of correctly predicted positive outcomes out of all predicted positive outcomes.
  Sensitivity (True Positive Rate, TPR): The proportion of actual positive outcomes that are correctly identified by the model.
  Specificity (True Negative Rate, TNR): The proportion of actual negative outcomes that are correctly identified by the model.

SUMMARY:
PROSAH-MPC, a collaborative research project among neurosurgical centers in China, focuses on aneurysmal subarachnoid hemorrhage (aSAH). Its aim is to identify prognostic factors and develop robust prediction models for complications, disability, and mortality in aSAH patients. By leveraging a large, multi-center, prospective cohort design, PROSAH-MPC aims to overcome limitations of past studies and provide a more comprehensive understanding of the disease.

DETAILED DESCRIPTION:
PROSAH-MPC (Prognostic Factors and Prediction Models in Aneurysmal Subarachnoid Hemorrhage Multi-Center Prospective Cohort) is an ambitious research endeavor that brings together a consortium of neurosurgical centers across various regions to comprehensively investigate the complexities of aneurysmal subarachnoid hemorrhage (aSAH). This multi-faceted study aims to unlock the prognostic factors that underpin the outcomes of patients afflicted with this severe and often life-threatening cerebrovascular disorder.

The primary objective of PROSAH-MPC is to construct and validate robust prediction models that can accurately forecast the risks of complications, disability, and mortality in aSAH patients. By leveraging the strengths of a large, multi-center, prospective cohort design, the study aims to overcome the limitations of previous single-center, limited sample size, or retrospective studies, enabling a more holistic and generalizable understanding of the disease.

Central to the study is the collection of extensive clinical and radiological data from enrolled patients, including demographics, medical histories, treatment regimens, radiological features, and follow-up outcomes. Radiomic analysis of imaging data, such as CT and MRI scans, will be employed to extract subtle but crucial features that may predict patient outcomes by deep learning. This data-rich approach ensures that the prediction models are built on a solid foundation of evidence-based knowledge.

PROSAH-MPC's ultimate goal is to transform the way we approach aSAH management by providing clinicians with reliable tools to assess individual patient risks and tailor treatment plans accordingly. The validated prediction models have the potential to enhance early recognition of high-risk patients, facilitate timely interventions, and ultimately improve patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage confirmed by computed tomography (CT);
* Cerebral angiography (CTA) and digital subtraction angiography (DSA) examination confirming intracranial aneurysm rupture as the cause of the subarachnoid hemorrhage;
* Blood routine, biochemical function, blood coagulation function, and craniocerebral CT performed within 24 hours of symptom onset;
* Underwent aneurysm clipping by surgery or endovascular embolization within 72 hours after-onset.

Exclusion Criteria:

* Aneurysm rupture bleeding time exceeding 24 hours before hospital admission;
* Incomplete image data or blood test information;
* Long-term use of anticoagulant medications such as aspirin or warfarin;
* Admitted to hospital with active infectious diseases;
* long-term anticoagulant drugs such as aspirin, wave dimensions;
* Presence of other intracranial vascular malformations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Aneurysmal Subarachnoid Hemorrhage (aSAH)
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) for evaluating the prognosis | 12 months post-event
  A score of 3 or greater on the mRS indicates a poor prognosis, with significant disability or dependence on others for daily activities.
  A score less than 3 indicates a good prognosis, with the patient being able to live independently with minimal or no disability.
Delayed cerebral ischemia (DCI) | 30 days post-event
  DCI is a common complication after aSAH and refers to a decline in neurological status or the presence of new infarctions on imaging, typically occurring days to weeks after the initial hemorrhage.

SECONDARY OUTCOMES:
Rebleeding | 30 days post-event
  This outcome measures the occurrence of recurrent intracranial hemorrhage from the same or another aneurysm within the study period.
Intracranial Aneurysm Re-Rupture | 30 days post-event
  This refers to the re-rupture of the aneurysm that caused the initial aSAH or the rupture of a different aneurysm.
Hydrocephalus | 30 days post-event
  Hydrocephalus is the abnormal accumulation of cerebrospinal fluid in the brain's ventricles, leading to their dilation.
Clearing Rate of Subarachnoid Hemorrhage | 14 days post-admission CT scan
  This outcome measures the reduction in the volume of subarachnoid hemorrhage over time, quantified using BrainHemoAI software by comparing admission CT scans to subsequent scans (e.g., at discharge or follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Xingen Zhu, Prof, Study Chair — Second Affiliated Hospital of Nanchang University; Qianxue Chen, Prof, Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Du S, Wu Y, Tao J, Shu L, Yan T, Xiao B, Lv S, Ye M, Gong Y, Zhu X, Hu P, Wu M. Development and Validation of Machine Learning Models for Outcome Prediction in Patients with Poor-Grade Aneurysmal Subarachnoid Hemorrhage Following Endovascular Treatment. Ther Clin Risk Manag. 2025 Mar 7;21:293-307. doi: 10.2147/TCRM.S504745. eCollection 2025. PMID 40071129
- [Derived] Shu L, Xiao B, Jiang Y, Tang S, Yan T, Wu Y, Wu M, Lv S, Lai X, Zhu X, Hu P, Ye M. Comparison of LVIS and Enterprise stent-assisted coiling embolization for ruptured intracranial aneurysms: a propensity score-matched cohort study. Neurosurg Rev. 2024 Sep 7;47(1):560. doi: 10.1007/s10143-024-02756-8. PMID 39242449